CLINICAL TRIAL: NCT05912998
Title: Comparative Study Between Autologous Adipose Tissue Graft With Hyaline Catilage Versus Microfracture for Treatment of Articular Cartilage Defects
Brief Title: Comparative Study Between Autologous Adipose Tissue Graft Versus Microfracture for Treatment of Articular Cartilage Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelgaliel Mohamed, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGMM
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cartilage regeneration (Active Comparator): 35 patient will have knee arthroscopy and cartilage regeneration technique and high tibial osteotomy
  Interventions: Procedure: cartilage regeneration technique
- microfracture (Active Comparator): 35 patient will have knee arthroscopy and microfracture with high tibial osteotomy
  Interventions: Procedure: cartilage regeneration technique
- high tibial osteotomy (Placebo Comparator): 35 patient will have knee arthroscopy and high tibial osteotomy
  Interventions: Procedure: cartilage regeneration technique

INTERVENTIONS:
Procedure: cartilage regeneration technique — autologous adipose tissue graft with hyaline cartilage graft mixed with fiberinglu

SUMMARY:
Knee arthroscopy using standard portals will be performed in three groups. Complete evaluation of all intra -articular structures will be performed followed by accurate localization of the cartilage defect and measurement of its dimensions. The cartilage lesion grading according to the International Cartilage Repair Society system (ICRS). The patients assigned for the first group will have Liposuction through a minor 1 cm incision on the abdomen to obtain adequate amount of emulsified adipose tissues (50 - 60 cc). Autologous adipose tissue will be mixed with autologous hyaline cartilage obtained from non-weight bearing areas of the knee in prepared mold. The graft will be mixed with fibrin glue and left to solidify a little. After obtaining the fashioned graft from the mold it will be fixed in to the defect site by fibrin glue through mini open approach and stability of the implant fitted in the site will evaluated by gentle cycling of the joint. During the graft preparation, a high tibial osteotomy will be performed. Patients assigned for the second group will have microfracture in association with open wedge high tibial osteotomy. Patients assigned for the third group will have open wedge high tibial osteotomy. Standard titanium T locked plate will be used to fix the open wedge osteotomy in the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18 to 60 years old.
* Cartilage defect size range 2-5 cm2.
* Outer Bridge classification II & III.
* Single full thickness symptomatic femoral condyles ulcer.
* Varus deformity of the affected knee 50 - 100.

Exclusion Criteria:

* Advanced knee osteoarthritis.
* Knee range of motion less than 1000.
* Ligamentous injury of the affected knee.
* Recent intra articular injection of any type with in last 6 months.
* Fracture around the knee.
* Inflammatory joints disorders.
* Tumors.
* Immunocompromised patients.
* Body mass index < 35
* Valgus deformed knee any degree
* Sever varus deformed knee < 10 0

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of International Knee Documentation Committee (IKDC) scores | one year